CLINICAL TRIAL: NCT06493734
Title: Stereotactic Body Radiation Therapy After Chemotherapy for Unresectable Perihilar Cholangiocarcinoma: A Multicenter Phase II Trial (The STRONG 2 Trial)
Brief Title: Stereotactic Body Radiation Therapy After Chemotherapy for Unresectable Perihilar Cholangiocarcinoma
Acronym: STRONG II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86210.078.24
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-12

CONDITIONS: Klatskin Tumor
Keywords: Klatskin tumor; Perihilar cholangiocarcinoma; Stereotactic body radiation therapy
MeSH Terms: conditions — Klatskin Tumor | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic body radiation therapy (Experimental): Single-arm study
  Interventions: Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — SBRT will be delivered in 15 fractions of 4 to 4.5Gy (risk-adapted), one fraction each weekday for 3 weeks.

SUMMARY:
The objective of this study is to evaluate the efficacy of stereotactic body radiation therapy (SBRT) as additional treatment after standard chemotherapy regarding tumor local control, toxicity, progression-free survival (PFS), overall survival and quality of life. In addition, the objective is to explore the value of immunodynamics in peripheral blood for predicting PFS in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Rationale:

For patients with perihilar cholangiocarcinoma, surgery is the only treatment modality that can result in cure. Unfortunately, in the majority of these patients the tumors are found to be unresectable at presentation due to local invasive tumor growth or the presence of distal metastases. For patients with unresectable cholangiocarcinoma, palliative chemotherapy is the standard treatment, yielding an estimated median overall survival of 12-15.2 months.

There is no evidence from randomized trials that support the routine use of stereotactic body radiation therapy (SBRT) for cholangiocarcinoma. The STRONG phase I feasibility study showed favorable outcomes regarding safety, and the therapy was generally well tolerated. Based upon these observations, a phase II multi-center study with SBRT after chemotherapy in patients with unresectable perihilar cholangiocarcinoma is proposed, in order to further research the efficacy of adding SBRT to standard chemotherapy.

In addition, an explorative translational research component is part of the study, in which peripheral immunodynamics, specifically myeloid nuclear factor kappa-light-chain enhancer of activated B cells (NF-kB) signaling and interferon-stimulated genes (ISG) responses within the myeloid cells, may help to predict survival after chemotherapy and may also help to predict the value of additional treatment with radiotherapy.

Objective:

The objective of this study is to evaluate the efficacy of SBRT as additional treatment after standard chemotherapy regarding tumor local control, toxicity, progression-free survival (PFS), overall survival and quality of life. In addition, to explore the value of immunodynamics in peripheral blood for predicting PFS in patients undergoing chemotherapy.

Study design:

Single-arm, multicenter phase II study.

Study population:

The initial translational part of the study will be performed in patients diagnosed with unresectable perihilar cholangiocarcinoma, 18 years of age or older, T1-4 N0-2 M0 (AJCC staging 8th edition), eligible for gemcitabine-based chemotherapy. Exclusion criteria are tumor extension into either stomach, colon, duodenum, pancreas or abdominal wall. After completion of chemotherapy and no local or distant progression during or after chemotherapy, the patients will proceed to SBRT if they are still eligible based on the inclusion and exclusion criteria. It may occur that patients do not give consent for the translational part of the study, but they may wish to participate in the SBRT part of the trial and vice versa. Sample size will be 30 patients.

Intervention:

SBRT will be delivered in 15 fractions of 4 to 4.5Gy after 8 cycles of chemotherapy. In case of toxicity causing premature termination of systemic treatment, the patient can still proceed to SBRT.

Main study parameters/endpoints:

The primary endpoint of this study is local tumour control, defined as time from inclusion to local radiological progression. Definition of progression is based on response evaluation criteria in solid tumours (RECIST) 1.1.

Secondary endpoints:

* Toxicity according to the Common Toxicity Criteria for Adverse Events (CTCAE) V.5.0 grading system.
* Biliary stent-related events (SRE).
* Progression-free survival defined as time from inclusion until radiological progression. Definition of progression is based on RECIST 1.1.
* Overall survival defined as time from inclusion until death from any cause.
* Quality of life (QoL), assessed by means of the EuroQol (EQ)-5D-5L (measure of health outcome in general population), and the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 (QoL specific for patients with cancer) with the supplementary module EORTC QLQ-BIL21 (specific for CCA and gallbladder cancer).

ELIGIBILITY:
Inclusion criteria translational part of the study:

In order to be eligible to participate in the translational part of the study, a subject must be discussed in a liver tumor board, should be eligible for gemcitabine-based chemotherapy (and immunotherapy, if applicable), and should meet all of the following criteria pre-chemotherapy:

* Perihilar cholangiocarcinoma (pCCA) according to the criteria of the Mayo Clinic, Rochester: a positive or strongly suspicious intraluminal brush cytology or biopsy, or a radiographic malignant appearing stricture plus either: CA 19-9>100 U/ml in the absence of acute bacterial cholangitis, or polysomy on fluorescence in situ hybridization (FISH), or a well-defined mass on cross sectional imaging
* One tumor mass
* Unresectable tumor or patient deemed unfit for surgery
* T1-T4 (AJCC staging 8th edition), N0-N2-M0 (AJCC staging 8th edition), radiologically or pathologically suspect. N1 is defined as one to three affected lymph nodes typically involving the hilar, cystic duct, common bile duct, hepatic artery, posterior pancreatoduodenal, and portal vein lymph nodes. N2 is defined as four or more affected lymph nodes from the sites described for N1. Endoscopic ultrasound (EUS) is leading in identifying pathological lymph nodes compared to CT.
* In case of (underlying) liver cirrhosis: Child-Pugh A
* Age ≥ 18 years
* ECOG performance status 0-1
* Written informed consent for the translational part of the study

Inclusion criteria SBRT part of the study:

In addition to the criteria mentioned above, patients should meet the following criteria to be eligible for the treatment with SBRT:

* Measurable disease to be selected as a target on a computed tomography (CT) or magnetic resonance imaging (MRI) scan, according to RECIST 1.1 criteria
* Finished gemcitabine-based chemotherapy treatment, preferably 8 cycles. If less cycles are given, patients are still eligible for this study
* Bilirubin ≤3.0 times normal value, aspartate aminotransferase (AST)/alanine transaminase (ALT) ≤5 times ULN
* Platelets ≥ 50x10E9/ l, Leukocytes > 1.5x10E9/l, Hemoglobin (Hb) > 6 mmol/l
* Willing and able to comply to the follow-up schedule
* Able to start SBRT within 12 weeks after completion of chemotherapy and immuno-therapy (if applicable)
* Written informed consent for the SBRT part of the study

Exclusion criteria translational part of the study:

* Prior surgery or transplantation of the liver
* Tumor extension in stomach, colon, duodenum, pancreas or abdominal wall
* Ascites
* Prior radiotherapy to the liver
* Current pregnancy
* Affected lymph nodes outside the regions described in the inclusion criteria

Exclusion criteria SBRT part of the study:

Progression (local or distant) during or after chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Local tumor control | 42 months (maximum follow-up time)
  Local tumor control is defined as time from inclusion to local radiological progression. Definition of progression is based on response evaluation criteria in solid tumors (RECIST) 1.1. In RECIST 1.1, response of a tumor to treatment is defined as either complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 42 months (maximum follow-up time)
  PFS is defined as time from inclusion until radiological progression. Definition of progression is based on RECIST 1.1.
Overall survival (OS) | 42 months (maximum follow-up time)
  OS is defined as time from inclusion until death from any cause.
Adverse events | 42 months (maximum follow-up time)
  Adverse events assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) V.5.0
Biliary stent-related events (SRE) | 42 months (maximum follow-up time)
  The definition of SRE in this study is based on the definition used in the study by Lamarca et al. (https://doi.org/10.3748/wjg.v22.i26.6065). A SRE is defined as any one or more of the following: 1. any episode of jaundice which is considered significant enough for new stenting or medical treatment and is confirmed by radiological imaging to be associated with biliary dilatation; 2. any episode of infection which is clinically in keeping with cholangitis (bile duct infection) requiring antibiotic therapy; 3. bacteraemia with isolation in blood cultures of bacteria suspected to have originated in the biliary tract; and 4. any episode of cholecystitis or gallbladder perforation.
Quality of life (QoL) - EQ-5D-5L | 36 months
  Assessed by means of the EuroQol (EQ)-5D-5L (measure of health outcome in general population).
Quality of life (QoL) - QLQ-C30 | 36 months
  Assessed by means of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 (QoL specific for patients with cancer).
Quality of life (QoL) - QLQ-BIL21 | 36 months
  Assessed by means of the supplementary module EORTC QLQ-BIL21 (specific for CCA and gallbladder cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Méndez Romero, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- Belgium (2):
  - Antwerp University Hospital / Sint-Augustinus Gasthuiszusters, Wilrijk, Antwerp
  - University Hospital Brussels / Jules Bordet Institute, Brussels, Brussels Capital
- Netherlands (6):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center+ / Maastro Clinic Maastricht, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Erasmus MC, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Loosbroek SY, Milder MTW, de Ruysscher D, Vaes RDW, den Toom W, Willemssen F, Eskens F, Homs MYV, Groot Koerkamp B, van Driel LMJW, Seppenwoolde Y, van Werkhoven E, Intven M, Haj Mohammad N, de Bruijne J, Versteijne E, Bruynzeel AM, Brandts F, Erdmann JI, Westdorp H, Braam PM, Tjwa ETTL, Bouchart C, Demols A, Gulyban A, Buijsen J, de Vos-Geelen J, Dewulf M, Joye I, Vandamme T, Vonghia L, de Groot DJ, Dieters M, Ubbels FJF, Hoogwater FJH, Heijmen B, Mendez Romero A PHD. STRONG II trial: stereotactic body radiation therapy following chemotherapy for unresectable perihilar cholangiocarcinoma - a single-arm multicentre phase II study. BMJ Open. 2025 Jul 16;15(7):e097545. doi: 10.1136/bmjopen-2024-097545. PMID 40669914